CLINICAL TRIAL: NCT04769765
Title: Evaluation of the Feasability of a Care Pathway Integrating Collaborative Tele-expertise for the Prevention of Recurrent Hospitalisations for Patients With Diabetes
Brief Title: Feasability of a Care Pathway Integrating Collaborative Tele-expertise to Prevent Recurring Hospitalisations for Diabetic Patients
Acronym: TELXCODIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: * Low involvement of required centers despite positive responses to feasibility surveys
  * Lack of people available for each visio (2 to 3 centers present at most out of the 8 planned)
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Montpellier (Other); Alès Hospital (Unknown); Bagnols sur Cèze Hospital (Unknown); Sète Hospital (Unknown); Narbonne Hospital (Other); Béziers Hospital (Unknown); Centre hospitalier de Perpignan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ARS/2018/AMG-01
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Establishment of a care pathway (basic and specific) discussed and validated via a tele-expertise pluridisciplinary meeting by the 8 centers, quarterly monitoring of the course and for one year.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients on the basic diabetic program, eligible for an individualized care pathway. (Experimental): This research aims to demonstrate the feasibility of telemedicine through collaborative tele-expertise for the collegial definition of an individualized care pathway, in the context of diabetic patients with unscheduled hospitalizations repeated throughout the year (≥ 2/year). The feasibility will be assessed by the number of patients who have had at least 3 of the 4 planned follow-up visits, that is to say, who are eligible for the individualized care pathway.
  Interventions: Other: Definition of the Individualized Care Pathway

INTERVENTIONS:
Other: Definition of the Individualized Care Pathway — Implementation of an individualized care pathway defined in concertation with a multidisciplinary tele-expertise meeting held every 3 months for one year. These multidisciplinary tele-expertise meetings will be held between each of the normal routine consultations which are part of the normal, basic diabetic program which includes a consultation with a dietitian, monitoring by a state-registered nurse and treatment prescribed by the patient's general practitioner (with or without a consultation with the clinical pharmacist).

SUMMARY:
Telemedicine for diabetic patients is currently based simply on remotely monitoring capillary blood glucose levels. This experimental approach remains limited to insulin-treated diabetic patients with sufficient motivation and ability to use connected devices and only considers one aspect of the care required by diabetic patients. So far, telemedicine has not offered a more global approach to the therapeutic support of patients. This failing leads to recurrent hospitalizations for acute metabolic events.

This project aims to demonstrate the feasibility of an individualized care pathway based on a multidisciplinary tele-medical network on a territorial scale. This pathway will include a base program with follow-up that can be adapted and revised thanks to the regular use of collaborative tele-expertise.

The possibility of monthly multidiciplinary meetings via Tele-expertise between the different diabetes centers of the hospital groups would help to define and implement an individualized care pathway for diabetic patients hospitalized on a recurring basis (≥2 hospitalizations/year), which would be defined collegially during the multidiciplinary meetings .

DETAILED DESCRIPTION:
Diabetes control, assessed on the level of glycated hemoglobin (HbA1c), improves complications such as microangiopathy. To reduce cardiovascular disease, better global management including an individualized care pathway is required. Inadequate care results in a high rate of re-hospitalizations during the year (approximately 15 to 20% of all diabetic patients).

So far, the only contribution of telemedicine in the context of diabetes has been the teletransmission of data from electronic monitoring logs, including insulin doses and capillary blood glucose measurements, to platforms accessible to healthcare teams (physicians and non-medical staff). Remote monitoring according to these methods can lead to asynchronous therapeutic proposals whose effectiveness on HbA1c levels has already been demonstrated and the contribution of telemonitoring has also already been validated on the improvement of certain cardiovascular risk factors.

However, this experimental approach remains limited to insulin-treated diabetic patients with sufficient capacity and motivation to use connected devices. It only considers one component of the care required by patients with diabetes.

Until now, telemedicine has not proposed a global approach to the therapeutic accompaniment of diabetic patients. Thus, recurrent hospitalizations for acute metabolic events (ketoacidosis, severe hypoglycemia) or complications related to diabetes (severe foot wounds, cardiovascular accidents, visual or renal alterations) are frequently observed.

The ambition of our project is therefore to demonstrate the feasibility of setting up an individualized care pathway that can be supported by a multidisciplinary tele-medical network on a regional level. This pathway will include a basic program and a follow-up which can be adapted and revised through regular use of collaborative tele-expertise.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients hospitalized on an unscheduled basis in the diabetology department of one of the 8 study centers.
* Patients with at least two unscheduled hospitalizations in less than one year (i.e. at least one other hospitalization in the last 365 days in addition to the hospitalization on the day of the pre-inclusion visit).
* Patient with diabetes for more than one year at the time of inclusion
* Patients affiliated to or beneficiary of a health insurance plan.

Exclusion Criteria:

* Patients with significant language barrier
* Homeless patients.
* Patients in a period of exclusion determined by another study.
* Minor patients.
* Patients under legal protection, guardianship or curatorship.
* Patient for whom it is impossible to give informed information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Number of patients eligible for the Individualized Care Pathway as well as the basic diabetic program. | At the end of the study period: Month 12 + 5 days
  After the intial pre-inclusion visit, 30 days before inclusion, a multidiciplinary tele-expertise meeting will be held to decide which patients are eligible for inclusion in the individualized care pathway. The aim is to demonstrate the feasibility of telemedicine through collaborative tele-expertise for the collegial definition of an individualized care pathway, in the context of diabetic patients with unscheduled hospitalization, iteratively over the year (≥ 2/year). The feasibility will be assessed by the number of inclusions and the number of patients included who have had at least 3 of the 4 planned follow-up visits.
Number of patients on the basic diabetic program, included in the study, who have completed at least three of the four scheduled follow-up visits. | At the end of the study period: Month 12 + 5 days
  This research aims to demonstrate the feasibility of telemedicine through collaborative tele-expertise for the collegial definition of an individualized care pathway, in the context of diabetic patients with unscheduled hospitalization, iteratively over the year (≥ 2/year). The feasibility will be assessed by :
  The number of inclusions and the number of patients included who have completed at least 3 of the 4 planned follow-up visits.

SECONDARY OUTCOMES:
Evolution of blood glucose (sugar) levels in patients benefitting from the individualized care pathway. | Month 0
  The rate of HbA1c will be measured as a percentage.
Evolution of blood glucose (sugar) levels in patients benefitting from the individualized care pathway. | Month 3
  The rate of HbA1c will be measured as a percentage.
Evolution of blood glucose (sugar) levels in patients benefitting from the individualized care pathway. | Month 6
  The rate of HbA1c will be measured as a percentage.
Evolution of blood glucose (sugar) levels in patients benefitting from the individualized care pathway. | Month 9
  The rate of HbA1c will be measured as a percentage.
Evolution of blood glucose (sugar) levels in patients benefitting from the individualized care pathway. | Month 12
  The rate of HbA1c will be measured as a percentage.
Re-hospitalization rate | 2 years (concernining the period M0 to M12)
  The SNIIRAM (Système National d'Information Inter Régimes de l'Assurance Maladie) which is the French Health Insurance database, will be used to observe the number of re-hospitalizations throughout the year. For each patient, in the database, YES or NO will be recorded to answer the question: Re-hospitalization? and, if the patient has been re-hospitalized, the number of re-hospitalizations will be noted.
Number of incidents of ketoacidosis | 2 years (Month -12 to Month 12)
  The number of serious incidents of ketoacidosis will be noted from data in the patient file.
Number of incidents of hypoglycemia | 2 years (Month -12 to Month 12)
  The number of serious incidents of hypoglygemia will be noted from data in the patient file.
Number of incidents of serious wounds | 2 years (Month -12 to Month 12)
  The number of serious wounds will be noted from data in the patient file.
Number of cardiovascular accidents | 2 years (Month -12 to Month 12)
  The number of cardiovascular accidents will be noted from data in the patient file.
Number of incidents of diabetic microangiopathy | 2 years (Month -12 to Month 12)
  The number of incidents of diabetic microangiopathy will be noted from data in the patient file.
Cost of care of diabetic patients | 2 years (Month -12 to Month 12)
  The total cost of caring for these diabetic patients who have had unscheduled hospitalization(s) during the year will be measured in Euros. Expenses will include consultations, hospitalizations, drug treatments, etc.). This information will be extracted from the French Health Insurance database (SNIIRAM).
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. Number of centers involved. | 1 year (Month 12)
  Number of centers involved in each multidisciplinary tele-expertise meeting.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise.Number of centers connected. | 1 year (Month 12)
  Number of centers connected at each multidisciplinary tele-expertise meeting.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise.Number of participants connected. | 1 year (Month 12)
  Number of participants per center connected at each multidisciplinary tele-expertise meeting.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. Duration of meetings. | 1 year (Month 12)
  Duration of each multidisciplinary tele-expertise meeting in terms of minutes.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise.Technical difficulties. | 1 year (Month 12)
  Number of technical difficulties encountered at each multidisciplinary tele-expertise meeting (connection etc.)
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. New patient files per center. | 1 year (Month 12)
  Number of new patient files presented per center.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. Patient follow-up files per center. | 1 year (Month 12)
  Number of patient follow-up files presented per center.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. New patient files at each meeting. | 1 year (Month 12)
  Number of new patient files presented at each multidisciplinary tele-expertise meeting.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. Patient follow-up files at each meeting. | 1 year (Month 12)
  Number of patient follow-up files presented at each multidisciplinary tele-expertise meeting.
Logistic feasability of managing these patients (who have had at least one unscheduled hospitalization during the year) by tele-expertise. Number of follow-up visits per patient per center. | 1 year (Month 12)
  Number of 3-monthly follow-up visits per patient per centre.

OTHER OUTCOMES:
Sex of patients | At the inclusion visit (Month 0)
  The sex of all patients' will be recorded (M/F/other).
Age of patients | At the inclusion visit (Month 0)
  All patients' ages will be recorded in years.
Weight of patients | At the inclusion visit (Month 0)
  All patients' weights will be recorded in kilograms.
Weight of patients | At the second visit (Month 3)
  All patients' weights will be recorded in kilograms.
Weight of patients | At the third visit (Month 6)
  All patients' weights will be recorded in kilograms.
Weight of patients | At the fourth visit (Month 9)
  All patients' weights will be recorded in kilograms.
Weight of patients | At the final visit (Month 12)
  All patients' weights will be recorded in kilograms.
Height of patients | At the inclusion visit (Month 0)
  All patients' heights will be recorded in centimeters.
Systolic blood pressure | At the inclusion visit (Month 0)
  Systolic blood pressure will be recorded for all patients in mmHg
Systolic blood pressure | At the second visit (Month 3)
  Systolic blood pressure will be recorded for all patients in mmHg
Systolic blood pressure | At the third visit (Month 6)
  Systolic blood pressure will be recorded for all patients in mmHg
Systolic blood pressure | At the fourth visit (Month 9)
  Systolic blood pressure will be recorded for all patients in mmHg
Systolic blood pressure | At the final visit (Month 12)
  Systolic blood pressure will be recorded for all patients in mmHg
Diastolic blood pressure | At the inclusion visit (Month 0)
  Diastolic blood pressure will be recorded for all patients in mmHg
Diastolic blood pressure | At the second visit (Month 3)
  Diastolic blood pressure will be recorded for all patients in mmHg
Diastolic blood pressure | At the third visit (Month 6)
  Diastolic blood pressure will be recorded for all patients in mmHg
Diastolic blood pressure | At the fourth visit (Month 9)
  Diastolic blood pressure will be recorded for all patients in mmHg
Diastolic blood pressure | At the final visit (Month 12)
  Diastolic blood pressure will be recorded for all patients in mmHg
Blood sugar levels | At the inclusion visit (Month 0)
  Blood sugar levels (HbA1c) will be recorded for all patients as a percentage
Blood sugar levels | At the second visit (Month 3)
  Blood sugar levels (HbA1c) will be recorded for all patients as a percentage
Blood sugar levels | At the third visit (Month 6)
  Blood sugar levels (HbA1c) will be recorded for all patients as a percentage
Blood sugar levels | At the fourth visit (Month 9)
  Blood sugar levels (HbA1c) will be recorded for all patients as a percentage
Blood sugar levels | At the final visit (Month 12)
  Blood sugar levels (HbA1c) will be recorded for all patients as a percentage
Glomerular Filtration Rate | At the inclusion visit (Month 0)
  Glomerular Filtration Rate will be recorded for all patients in ml/mn
Glomerular Filtration Rate | At the second visit (Month 3)
  Glomerular Filtration Rate will be recorded for all patients in ml/mn
Glomerular Filtration Rate | At the third visit (Month 6)
  Glomerular Filtration Rate will be recorded for all patients in ml/mn
Glomerular Filtration Rate | At the fourth visit (Month 9)
  Glomerular Filtration Rate will be recorded for all patients in ml/mn
Glomerular Filtration Rate | At the final visit (Month 12)
  Glomerular Filtration Rate will be recorded for all patients in ml/mn
Total cholesterol | At the inclusion visit (Month 0)
  Total cholesterol will be recorded for all patients in mmol/L
Total cholesterol | At the second visit (Month 3)
  Total cholesterol will be recorded for all patients in mmol/L
Total cholesterol | At the third visit (Month 6)
  Total cholesterol will be recorded for all patients in mmol/L
Total cholesterol | At the fourth visit (Month 9)
  Total cholesterol will be recorded for all patients in mmol/L
Total cholesterol | At the final visit (Month 12)
  Total cholesterol will be recorded for all patients in mmol/L
Low-density lipoprotein cholesterol | At the inclusion visit (Month 0)
  Low-density lipoprotein cholesterol will be recorded for all patients in mmol/L
Low-density lipoprotein cholesterol | At the second visit (Month 3)
  Low-density lipoprotein cholesterol will be recorded for all patients in mmol/L
Low-density lipoprotein cholesterol | At the third visit (Month 6)
  Low-density lipoprotein cholesterol will be recorded for all patients in mmol/L
Low-density lipoprotein cholesterol | At the fourth visit (Month 9)
  Low-density lipoprotein cholesterol will be recorded for all patients in mmol/L
Low-density lipoprotein cholesterol | At the final visit (Month 12)
  Low-density lipoprotein cholesterol will be recorded for all patients in mmol/L
High-density lipoprotein cholesterol | At the second visit (Month 0)
  High-density lipoprotein cholesterol will be recorded for all patients in mmol/L
High-density lipoprotein cholesterol | At the second visit (Month 3)
  High-density lipoprotein cholesterol will be recorded for all patients in mmol/L
High-density lipoprotein cholesterol | At the third visit (Month 6)
  High-density lipoprotein cholesterol will be recorded for all patients in mmol/L
High-density lipoprotein cholesterol | At the fourth visit (Month 9)
  High-density lipoprotein cholesterol will be recorded for all patients in mmol/L
High-density lipoprotein cholesterol | At the final visit (Month 12)
  High-density lipoprotein cholesterol will be recorded for all patients in mmol/L
Triglycerides | At the inclusion visit (Month 0)
  Triglycérides will be recorded for all patients in mmol/L
Triglycerides | At the second visit (Month 3)
  Triglycérides will be recorded for all patients in mmol/L
Triglycerides | At the third visit (Month 6)
  Triglycérides will be recorded for all patients in mmol/L
Triglycerides | At the fourth visit (Month 9)
  Triglycérides will be recorded for all patients in mmol/L
Triglycerides | At the final visit (Month 12)
  Triglycérides will be recorded for all patients in mmol/L
Treatment method | At the inclusion visit (Month 0)
  The treatment method will be recorded for all patients : injection or pump, non-insulin antidiabetics, basal or multi-injection insulin, oral anti-diabetic drugs; Dipeptidyl peptidase-4 inhibitor; glucagon-like peptide-1 analog, Statins, Beta-blockers, anti aggregation, Antibiotics: (YES/NO).
Treatment method | At the second visit (Month 3)
  The treatment method will be recorded for all patients : injection or pump, non-insulin antidiabetics, basal or multi-injection insulin, oral anti-diabetic drugs; Dipeptidyl peptidase-4 inhibitor; glucagon-like peptide-1 analog, Statins, Beta-blockers, anti aggregation, Antibiotics: (YES/NO).
Treatment method | At the third visit (Month 6)
  The treatment method will be recorded for all patients : injection or pump, non-insulin antidiabetics, basal or multi-injection insulin, oral anti-diabetic drugs; Dipeptidyl peptidase-4 inhibitor; glucagon-like peptide-1 analog, Statins, Beta-blockers, anti aggregation, Antibiotics: (YES/NO).
Treatment method | At the fourth visit (Month 9)
  The treatment method will be recorded for all patients : injection or pump, non-insulin antidiabetics, basal or multi-injection insulin, oral anti-diabetic drugs; Dipeptidyl peptidase-4 inhibitor; glucagon-like peptide-1 analog, Statins, Beta-blockers, anti aggregation, Antibiotics: (YES/NO).
Treatment method | At the final visit (Month 12)
  The treatment method will be recorded for all patients : injection or pump, non-insulin antidiabetics, basal or multi-injection insulin, oral anti-diabetic drugs; Dipeptidyl peptidase-4 inhibitor; glucagon-like peptide-1 analog, Statins, Beta-blockers, anti aggregation, Antibiotics: (YES/NO).
Date of diagnosis of diabetes | At the inclusion visit (Month 0)
  For each patient, the date and the year when diabètes was first diagnosed will be recorded.
Complications | At the inclusion visit (Month 0)
  The presence of any eventual complications will be noted for each patient : nephropathy, retinopathy, coronaropathy, trophic disorders, coma (YES/NO)
Complications | At the second visit (Month 3)
  The presence of any eventual complications will be noted for each patient : nephropathy, retinopathy, coronaropathy, trophic disorders, coma (YES/NO)
Complications | At the third visit (Month 6)
  The presence of any eventual complications will be noted for each patient : nephropathy, retinopathy, coronaropathy, trophic disorders, coma (YES/NO)
Complications | At the fourth visit (Month 9)
  The presence of any eventual complications will be noted for each patient : nephropathy, retinopathy, coronaropathy, trophic disorders, coma (YES/NO)
Complications | At the final visit (Month 12)
  The presence of any eventual complications will be noted for each patient : nephropathy, retinopathy, coronaropathy, trophic disorders, coma (YES/NO)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Centre Hospitalier d'Alès, Alès
  - CH de Bagnols sur Cèze, Bagnols-sur-Cèze
  - CH de Beziers, Béziers
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CH de Narbonne HÔTEL DIEU, Narbonne
  - Centre Hospitalier Saint Jean, Perpignan
  - Hopital St Clair Hbt Sete, Sète